CLINICAL TRIAL: NCT06404385
Title: Prospective Clinical Study on the Accuracy of Static Computer-assisted Implant Surgery in Patients Rehabilitated With Distal Free-end Implants. Conventional Versus CAD-CAM Surgical Guides
Brief Title: Accuracy of Static Computer-assisted Implant Surgery in Distal Free-end Scenarios
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Berta García Mira, Assistant Professor of Stomatology, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: H20190402125847
Record Dates: First submitted 2024-04-29; First posted 2024-05-08 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Dental Implant; Computer-assisted
Keywords: accuracy; computer-assisted surgery; computer-aided design; analogic; dental implants

STUDY DESIGN:
Intervention Model Description: A prospective, controlled, examiner- and statistician-blinded, parallel-arm quasi-experimental study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional surgical guide (Active Comparator): Implants (Straumann®) placed with an analogic laboratory surgical guide
  Interventions: Procedure: Static computer-assisted guided surgery with analogic guide
- Computer aided design - computer aided manufacturing (CAD-CAM) surgical guide (Experimental): Implants (Straumann®) placed with static computer-assisted implant surgery
  Interventions: Procedure: Static computer-assisted guided surgery with CAD-CAM surgical guide

INTERVENTIONS:
Procedure: Static computer-assisted guided surgery with analogic guide — coDiagnostix9® planning software
  Other Names: Conventional laboratory surgical guide; gonyX®
  Arms: Conventional surgical guide
Procedure: Static computer-assisted guided surgery with CAD-CAM surgical guide — coDiagnostix9® planning software
  Other Names: CAD-CAM surgical guide
  Arms: Computer aided design - computer aided manufacturing (CAD-CAM) surgical guide

SUMMARY:
Technological advances have influenced the approach to implant treatment. One of the fields presently experiencing rapid development is static computer-assisted guided surgery (sCAIS), which allows transfer of the virtual implant planning to the mouth of the patient, based on the use of a surgical guide. In sCAIS there is a deviation between the virtually planned implant position and the actual position of the implant placed during surgery. A recent review analyzed only fully guided implants and recorded a mean coronal horizontal deviation (CHD) of 1.12 mm (standard deviation [SD] = 0.08), a mean apical horizontal deviation (AHD) of 1.41 mm (SD = 0.1), a mean vertical deviation (VD) of 0.12 mm (SD = 0.23), and a mean angular deviation (AD) of 3.58º (SD = 0.2).

The aim of the present study was to compare the accuracy of CAD-CAM and conventional guides in candidates for distal free-end implant treatment, and to analyze the effects of possible confounding factors inherent to the patient or the surgical technique employed.A prospective, controlled and blinded quasi-experimental study was carried out involving 27 patients with 76 implants distributed into two groups according to the surgical guide manufacturing approach used: conventional (control group [CG]) or CAD-CAM (test group [TG]). The implants were planned virtually with the planning software, and the surgical guides were manufactured. Fully guided implant placement was carried out, and the deviations were measured along with other secondary variables as potential confounding factors.

DETAILED DESCRIPTION:
Planning of the implants is made in the ideal prosthetic position based on a previous CAD-CAM (computer aided design - computer aided manufacturing) wax-up. sCAIS facilitates correct prosthetic emergence and therefore contributes to secure optimum esthetic and biological outcomes, affording long-term stability of the soft and hard tissues.

These surgical guides can be manufactured using CAD-CAM or conventional technologies in the laboratory, employing drilling machines or mechanical positioners. In the case of the conventional guide manufactured in the laboratory, the technician creates a radiological guide that is then converted into a surgical guide - the whole process being analogic, except for planning of the implants. At present, and with the development of digital workflows, CAD-CAM procedures are used for both the design and manufacture of the surgical guide, using different processes. This simplifies the workflow, which can reduce the costs of smaller rehabilitations.

Clinical studies on accuracy published in the literature are heterogeneous, with differences in the systems used, the surgical technique, the type of surgical guide support or the type of edentulism involved.These data justify further research in humans, focusing on fully sCAIS, in order to reduce heterogeneity. Furthermore, a review of the literature revealed a lack of clinical publications on the accuracy of CAD-CAM surgical guides compared to conventional guides. Therefore, the aim of the present study was to compare the accuracy of CAD-CAM and conventional guides in candidates for distal free-end implant treatment, and to analyze the effects of possible confounding factors inherent to the patient or the surgical technique employed. Intra- and postoperative complications of the surgical technique were also evaluated, as well as implant success and peri-implant marginal bone loss. Hence, the null hypothesis of the study was the absence of any difference in accuracy between both guides.

A prospective, controlled, examiner- and statistician-blinded, parallel-arm quasi-experimental study was carried out at the University of Valencia (Valencia, Spain). Two groups were established according to the surgical guide design involved: conventional (control group [CG]) or CAD-CAM (test group [TG]).

ELIGIBILITY:
Inclusion Criteria:

* Indication of fixed prosthesis over at least two consecutive implants.
* Sufficient residual crest for placing at least two implants 4.1 mm in diameter and 8 mm in length.
* Mature bone and healthy soft tissues.
* Implants placed via fully guided surgery.
* Age > 18 years.
* Good general health.
* Non-smokers or smokers of < 10 cigarettes/day (pipe smokers excluded).
* Oral hygiene index < 3 and bleeding index < 25%.
* Pre- and post- CBCT scan for analysis of accuracy.
* Periapical radiographs at loading and after one year.

Exclusion Criteria:

* Contraindications to implant therapy
* Locations with acute infection.
* Pregnant or nursing women.
* Lack of follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-09-11 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Accuracy in implants: vertical, apical and coronal horizontal deviations | 1 week post-operative
  New CBCT scans were obtained in all patients after implant placement . The coDiagnostix9® application was used to match the pre- and postoperative CBCT images and to compare the axis positions of the planned and placed implants. The vertical, apical and coronal horizontal deviations in millimeters (VD, AHD and CHD), were recorded between the long axis of the virtual planned and actual placed implant. Measured in millimeters
Accuracy in implants: angular deviation | 1 weel post-operatiive
  New CBCT scans were obtained in all patients after implant placement . The coDiagnostix9® application was used to match the pre- and postoperative CBCT images and to compare the axis positions of the planned and placed implants. The angular deviation in degrees (AD), was recorded between the long axis of the virtual planned and actual placed implant. Measured in degrees.

SECONDARY OUTCOMES:
Intraoperative complications | Intra-operative
  Surgical guide fitting, retention, drill access, guide fracture, I
Postoperative complications | One month after implant placement
  Infection, bleeding, edema, neurological alterations, pain, swelling
Implant success | One year of implant loading
  Success is defined as no permanent peri implant radiographic translucency, no sign of peri-implant infection with putrid secretion, absence of persistent pain, dysesthesia, and/or foreign-body feeling
Peri-implant marginal bone loss | One year of implant loading
  Radiographic assessment of the marginal bone loss around the implants

CONTACTS AND LOCATIONS:
Overall Officials: MIGUEL PEÑARROCHA-DIAGO, Phd, DDS, Study Director — University of Valencia
Locations (1):
- University of Valencia. Faculty of Medecine and Dentistry. CLINICA ODONTOLOGICA, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
Patients' personal data will not be published, however, the results of the scientific study will be published in a scientific dental journal.

REFERENCES:
- [Background] Balaguer-Marti JC, Canet-Lopez A, Penarrocha-Diago M, Romeo-Rubio M, Penarrocha-Diago M, Garcia-Mira B. Influence of Splint Support on the Precision of Static Totally Guided Dental Implant Surgery: A Systematic Review and Network Meta-analysis. Int J Oral Maxillofac Implants. 2023 Jan-Feb;38(1):157-168. doi: 10.11607/jomi.9796. PMID 37099571
- [Background] Bover-Ramos F, Vina-Almunia J, Cervera-Ballester J, Penarrocha-Diago M, Garcia-Mira B. Accuracy of Implant Placement with Computer-Guided Surgery: A Systematic Review and Meta-Analysis Comparing Cadaver, Clinical, and In Vitro Studies. Int J Oral Maxillofac Implants. 2018 January/February;33(1):101-115. doi: 10.11607/jomi.5556. Epub 2017 Jun 20. PMID 28632253
- [Background] Chen X, Yang Z, Wang Y, Fu G. Fixation Pins Increase the Accuracy of Implant Surgery in Free-End Models: An In Vitro Study. J Oral Maxillofac Surg. 2023 May;81(5):593-601. doi: 10.1016/j.joms.2022.12.017. Epub 2023 Jan 28. PMID 36716792
- [Background] El Kholy K, Lazarin R, Janner SFM, Faerber K, Buser R, Buser D. Influence of surgical guide support and implant site location on accuracy of static Computer-Assisted Implant Surgery. Clin Oral Implants Res. 2019 Nov;30(11):1067-1075. doi: 10.1111/clr.13520. Epub 2019 Aug 20. PMID 31381178
- [Background] El Kholy K, Janner SFM, Schimmel M, Buser D. The influence of guided sleeve height, drilling distance, and drilling key length on the accuracy of static Computer-Assisted Implant Surgery. Clin Implant Dent Relat Res. 2019 Feb;21(1):101-107. doi: 10.1111/cid.12705. Epub 2018 Dec 27. PMID 30589502
- [Background] Kessler A, Le V, Folwaczny M. Influence of the tooth position, guided sleeve height, supporting length, manufacturing methods, and resin E-modulus on the in vitro accuracy of surgical implant guides in a free-end situation. Clin Oral Implants Res. 2021 Sep;32(9):1097-1104. doi: 10.1111/clr.13804. Epub 2021 Jul 17. PMID 34218450
- [Background] Khorsandi D, Fahimipour A, Abasian P, Saber SS, Seyedi M, Ghanavati S, Ahmad A, De Stephanis AA, Taghavinezhaddilami F, Leonova A, Mohammadinejad R, Shabani M, Mazzolai B, Mattoli V, Tay FR, Makvandi P. 3D and 4D printing in dentistry and maxillofacial surgery: Printing techniques, materials, and applications. Acta Biomater. 2021 Mar 1;122:26-49. doi: 10.1016/j.actbio.2020.12.044. Epub 2020 Dec 26. PMID 33359299
- [Background] Le V, Kessler A, Folwaczny M. Influence of DLP and SLA printer technology on the accuracy of surgical guides for implant dentistry in free-end situations. Int J Comput Dent. 2023 Sep 26;26(3):217-226. doi: 10.3290/j.ijcd.b3774115. PMID 36625374
- [Background] Matta RE, Bergauer B, Adler W, Wichmann M, Nickenig HJ. The impact of the fabrication method on the three-dimensional accuracy of an implant surgery template. J Craniomaxillofac Surg. 2017 Jun;45(6):804-808. doi: 10.1016/j.jcms.2017.02.015. Epub 2017 Feb 20. PMID 28363503
- [Background] Putra RH, Yoda N, Astuti ER, Sasaki K. The accuracy of implant placement with computer-guided surgery in partially edentulous patients and possible influencing factors: A systematic review and meta-analysis. J Prosthodont Res. 2022 Jan 11;66(1):29-39. doi: 10.2186/jpr.JPR_D_20_00184. Epub 2021 Jan 26. PMID 33504723
- [Derived] Berta GM, Luigi C, Miguel PD, Carlos BJ. Prospective Clinical Study on the Accuracy of Static Computer-Assisted Implant Surgery in Patients With Distal Free-End Implants. Conventional Versus CAD-CAM Surgical Guides. Clin Oral Implants Res. 2025 Mar;36(3):314-324. doi: 10.1111/clr.14384. Epub 2024 Nov 23. PMID 39578942